CLINICAL TRIAL: NCT00294073
Title: Defining the Best Approach to Block the Pain After Knee Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEN#05-002; REC#02-030
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2005-08

CONDITIONS: Pain, Postoperative
Keywords: femoral block; fascia iliaca block; ACL repair; post-operative analgesia; knee surgery; ACL damage; knee damage
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Procedure: Fascia Iliaca Block
Procedure: Femoral Block (with stimulating catheter)
Procedure: Femoral Block (without stimulating catheter)

SUMMARY:
The study aims to compare standard techniques used to control pain after knee surgery. The investigators hypothesize that the fascia iliaca block is faster, safer and as good as or better than the femoral block, with or without a stimulating catheter.

DETAILED DESCRIPTION:
60 patients being treated for ACL repair or knee arthroplasties under regional anesthesia will be randomized to three groups: Fascia Iliaca Block (FIB), Femoral Block (FB) with stimulating catheter or FB without stimulating catheter. A catheter will be placed according to each technique, before the surgery. A bolus of local anesthetic will be given pre-surgery and at the end of the operation, in all groups. A continuous infusion will be started for 48 hours. All patients receive a standard analgesia cocktail and rescue medication.

Pain and level of activity, as well as side effects, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming for ACL or knee prosthesis surgery
* Between 18-80 years old
* Consenting for spinal anesthesia

Exclusion Criteria:

* Major neurologic diseases
* Obesity with body mass index (BMI) > 30
* Infection at the punction sites (back and/or groin)
* Diabetes mellitus for longer than 5 years
* Coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
pain relief; measured by VAS at rest and on activity | before surgery, before discharge from PACU and on evenings of days 1, 2, 7, 60, 90
pain relief; measured by WOMAC | before surgery and at days 7, 60, 90
pain relief; evaluated from standard datasheet | over 48-hour period

SECONDARY OUTCOMES:
knee range of bending | measured before surgery, and at days 7, 60, 90
thigh circumference 20 cm above the knee | measured before surgery and at days 7, 60, 90
neurological exam of femorocutaneous, femoral and obturator nerves | evaluated once spinal anesthesia has worn off, post-surgery, before anesthesia
level of activity; measured using questionnaire | at 7-10 days and at 2 and 3 months
need for rescue analgesia | in recovery room and at home
need for second bolus or crossing over between groups

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Asenjo, MD, Principal Investigator — Montreal General Hospital
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Morau D, Lopez S, Biboulet P, Bernard N, Amar J, Capdevila X. Comparison of continuous 3-in-1 and fascia Iliaca compartment blocks for postoperative analgesia: feasibility, catheter migration, distribution of sensory block, and analgesic efficacy. Reg Anesth Pain Med. 2003 Jul-Aug;28(4):309-14. doi: 10.1016/s1098-7339(03)00183-4. PMID 12945024
- [Background] Salinas FV, Neal JM, Sueda LA, Kopacz DJ, Liu SS. Prospective comparison of continuous femoral nerve block with nonstimulating catheter placement versus stimulating catheter-guided perineural placement in volunteers. Reg Anesth Pain Med. 2004 May-Jun;29(3):212-20. doi: 10.1016/j.rapm.2004.02.009. PMID 15138905
- [Background] Williams BA, Kentor ML, Vogt MT, Vogt WB, Coley KC, Williams JP, Roberts MS, Chelly JE, Harner CD, Fu FH. Economics of nerve block pain management after anterior cruciate ligament reconstruction: potential hospital cost savings via associated postanesthesia care unit bypass and same-day discharge. Anesthesiology. 2004 Mar;100(3):697-706. doi: 10.1097/00000542-200403000-00034. PMID 15108988
- [Background] Eriksson E. Pain relief after ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2004 May;12(3):179. doi: 10.1007/s00167-004-0526-4. Epub 2004 Apr 21. No abstract available. PMID 15103457